CLINICAL TRIAL: NCT07341126
Title: Surveillance Digital Rectoscopy After Local Excision of Rectal Tumours
Brief Title: Use of a Novel Camera to Check the Bowel After Polyp or Tumour Removal
Acronym: R-ALERT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 363843
Record Dates: First submitted 2025-11-14; First posted 2026-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bowel Cancer; Polyp Rectal; Rectal Cancer; Rectal Adenocarcinoma; Rectal Adenoma
Keywords: LumenEye; Rectoscopy
MeSH Terms: conditions — Intestinal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Surveillance cohort: Patients undergoing surveillance following rectal tumour removal
  Interventions: Diagnostic Test: LumenEye X1 digital rectoscope

INTERVENTIONS:
Diagnostic Test: LumenEye X1 digital rectoscope — The LumenEye X1 is a novel digital rectoscope that introduces digital HD imaging and improved ergonomics to conventional rigid sigmoidoscopy.

SUMMARY:
1.1 Polyps or tumours in the lower part of the bowel (rectum) can be removed using instruments inserted through the bottom which avoids major surgery and the possibility of a stoma bag (colostomy). Afterwards, it is important to check the area with regular camera tests. If checks are delayed, re-growths could be serious and may be untreatable. COVID and other factors have led to long waiting lists for camera checks and in NHS Lothian around 20% of all camera checks are done more than 6 months late.

The investigators want to try a new camera and approach that would allow us to reduce waiting lists. Using a short camera called a 'rectoscope' to check the lower bowel has already been shown to be safe, comfortable and acceptable to patients with other conditions. In fact, patients are unlikely to feel or realise any difference between the rectoscope and standard camera tests.

The investigators want to show that this 'rectoscope' can be safely used in the outpatient clinic with an enema (suppository) instead of strong bowel medicine taken by mouth the day before. This would mean the camera checks happen on time and would reduce waiting lists for other important tests.

The investigators will include 30 patients across three stages of our study. In the first set of patients, the investigators will use the rectoscope alongside the usual endoscope in the endoscopy room using the usual oral bowel medicine. This stage will check the rectoscope is acceptable to the patient and the doctor. In the next 10 patients the investigators will use a suppository instead of oral bowel medicine still using both cameras. Finally, the investigators will use the rectoscope in the outpatient clinic with an suppository to show this is an easy, effective and acceptable way to deliver timely camera checks.

DETAILED DESCRIPTION:
BACKGROUND Transanal excision of rectal tumours describes the excision of both benign and malignant rectal lesions avoiding the need for major rectal resection. Traditional transanal approaches facilitated the excision of lower third rectal tumours using a trans-anal retractor. Since its introduction in the 1980s, transanal endoscopic microsurgery (TEMS) has established itself as an oncologically effective and safe approach to transanal excision of neoplasms throughout the rectum. More recent developments using laparoscopic (TAMIS) and now robotic platforms (R-TAMIS) provide alternative approaches. Local excision techniques are associated with reduced comorbidity when compared with radical rectal resection (i.e. Total Mesorectal Excision, TME) e.g. death, bleeding, genito-urinary dysfunction and anastomotic leak and need for a stoma. The development and evolution of neo-adjuvant therapy for rectal cancer with significant rates of complete response, demonstrates the potential for organ preservation and may be used alongside local excision techniques, as studied in the TREK, STAR-TREK and GRECCAR-2.

However, it is suggested that when performed for cancer, oncological outcomes may be poorer in patients undergoing local excision compared to radical resection. Current evidence regarding recurrence and survival rates is inconsistent, with some studies suggesting equivalent outcomes, but other studies reporting worse oncological outcomes. As such, regular, high quality post-operative surveillance of the rectum in patients under local excision is critical. Current methods of surveillance for the detection of recurrence commonly include multimodal radiological cross-sectional imaging (magnetic resonance imaging (MRI) and computerised tomography (CT)) and endoscopic (flexible sigmoidoscopy/colonoscopy) surveillance. There are currently no established UK guidelines for surveillance of this patient cohort, yet it is clear that even where local excision of a benign lesion is performed, endoscopic surveillance remains critical in identifying and managing recurrence or metachronous rectal pathology.

1.2 RATIONALE FOR STUDY

COVID-19 had a seismic impact on the provision of care across medicine, not least on the delivery of timely endoscopic examinations, resulting in a significant reduction in activity and exponential increase in waiting times which persists to date. Surveillance procedures are perhaps most at risk of delays, especially when triaged against patients with positive faecal immunohistochemistry tests (FIT) with a high chance of significant pathology. Local data indicates poor compliance with surveillance schedules (Table 1) particularly for endoscopic procedures. In total 20.8% of flexible sigmoidoscopy requests for surveillance after TEMS rectal cancer excision were performed 6 or more months after the scheduled time.

Year 1 2 3 Months 4 8 12 18 24 30 36 Total Number of Patients 36 34 34 33 32 32 32 Pelvic MRI 20 (56%) 15 (44%) 11 (32%) 10 (30%) 6 (19%) 5 (16%) 1 (3%) CT (CAP) 14 (41%) 8 (25%) 3 (9%) Flexible Sigmoidoscopy 15 (42%) 6 (18%) 8 (24%) 7 (21%) 2 (6%) 2 (6%) 2 (6%) Table 1 - Number (%) of Patients Receiving Surveillance <1 month from scheduled date

As such, alternative strategies for high quality direct visualisation of the rectum are required in such patients. Poor equipment and lack of bowel preparation currently precludes accurate surveillance in the outpatient setting in most UK institutions, unlike the 'office' set up in USA which frequently includes a endoscopy stack and enemas taken by the patient before clinic. LumenEye® X1 (SurgEase Innovations Ltd, London, UK) is a CE-marked digital rectoscope coupled to a telestration software platform, that enables high-definition rectal visualisation to be performed with the option of capture, storage and transfer of still or video rectal images taken during examination. Feasibility studies have been reported in both primary and secondary care. Early reports indicate high diagnostic yield coupled with low cost, suggesting that this device could provide safe and effective rectal surveillance while reducing demands on dedicated endoscopy units.

Alongside the clear potential to reduce burden on endoscopy services, the use of a digital rectoscope may provide attendant cost-savings and a reduction in morbidity associated with a reduction in bowel preparation use. The National Health Service best-practice tariff 2020/21 for diagnostic flexible sigmoidoscopy is £310 ($429) or £395 ($547) with biopsy, ignoring postage and laxative costs. The cost of the LumenEye® X1 system is estimated at approximately £50 ($69). The device and software license can be purchased for £20,000 ($27,600), and the disposables are between £30 and £50 ($41 and $69) depending on commitment and duration of contract. As such, there is the potential for a significant cost saving if digital rectoscopy in the outpatient clinic setting could replace flexible sigmoidoscopy in the endoscopy department for select indications. In NHS Lothian, standard bowel preparation for flexible sigmoidoscopy is sodium picosulfate. Therefore, the proposed use of rectoscopy provides an opportunity to reconsider the necessity for cleansing bowel preparation in patients needing rectal visualisation alone. Ignoring the cost alone, cleansing bowel preparation is inconvenient and associated with distress and potential medical risks. Such preparations can have a profound effect on the gut microbiome and metabolome, may cause abdominal pain, nausea, vomiting and risks fluid shifts and electrolyte derangements including severe symptomatic hyponatraemia.

The aim of the present study is firstly to assess the LumenEye® X1 digital rectoscope against traditional flexible sigmoidoscopy. Both procedures will be performed at the same appointment within the endoscopy suite. Comparative outcomes will include image quality, surgeon and patient tolerability. The null hypothesis is that there is no difference in image quality of tolerability between a standard flexible sigmoidoscopy and digital rectoscope. The second stage (stage 2) of the study will assess whether per rectum bowel preparation (glycerin suppository) is comparable to standard oral bowel cleansing in regards to quality of bowel preparation and visualisation of the rectum. The null hypothesis is that there is no difference in rectal visualisation between suppository and either of two oral bowel preparation regimes. In the final stage, participants requiring rectal surveillance (beyond their index site check) will be invited to attend outpatient clinic, with self-administered suppository in the department 30 minutes before the appointment. The participant will undergo digital rectoscopy in the outpatient ('office') room. The three-staged design ultimately aims to assess whether outpatient surveillance is safe, effective and tolerated using the LumenEye® X1 digital rectoscope in patients receiving per rectum bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

All participants who are capable of giving informed consent. All participants aged 16 years or over. All patients must have had a rectal tumour/ polyp removed within easy reach of the rigid sigmoidoscope.

All participants must be resident in the United Kingdom.

Exclusion Criteria:

Unable to give informed consent. Under the age of 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients must have had a rectal tumour/ polyp removed within easy reach of the rigid sigmoidoscope undergoing post-operative surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of diagnostic accuracy | Baseline
  LumenEye for the Detection of Rectal Pathology Including Tumour, Polyps and Inflammation. To provide pilot data within the small study for the diagnostic accuracy of the LumenEye system as compared to conventional flexible endoscopy.
  In the first 2 stages of the study LumenEye will be compared against flexible sigmoidoscopy. Sigmoidoscopy will be considered the gold standard and will be performed directly after the LumenEye procedure.
  Accuracy will be calculated in standard fashion based on observations of true / false positive/ negative observations alongside measures of sensitivity and specificity.

SECONDARY OUTCOMES:
Clinician Experience of LumenEye Examination | Baseline
  Assessing the the positive response rate by examining clinicians to their overall experience and certainty of diagnosis for each examination. Confidence in LumenEye findings and overall clinician experience will be measured using a standard 4-5 point likert scale.
Patient Experience of LumenEye Examination | Baseline
  Assessing the percentage of participants with positive responses to the patient experience questionnaire, which is answered with a 5 point Likert scale.
  Questions are as follows:
  The LumenEye examination was comfortable:
  Strongly disagree / Disagree / Neutral / Agree / Strongly agree
  If needed, I would be willing to undergo a further examination with a LumenEye in future Strongly disagree / Disagree / Neutral / Agree / Strongly agree
  What is your overall opinion of your experience with LumenEye assessment? Very poor / Poor / Neutral / Positive / Very positive
  The flexible sigmoidoscopy examination was comfortable:
  Strongly disagree / Disagree / Neutral / Agree / Strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Confidentiality

REFERENCES:
- [Background] Hyun JH, Alhanafy MK, Park HC, Park SM, Park SC, Sohn DK, Kim DW, Kang SB, Jeong SY, Park KJ, Oh JH. Initial local excision for clinical T1 rectal cancer showed comparable overall survival despite high local recurrence rate: a propensity-matched analysis. Ann Coloproctol. 2022 Apr;38(2):166-175. doi: 10.3393/ac.2021.00479.0068. Epub 2021 Oct 6. PMID 34610653
- [Background] Rullier E, Vendrely V, Asselineau J, Rouanet P, Tuech JJ, Valverde A, de Chaisemartin C, Rivoire M, Trilling B, Jafari M, Portier G, Meunier B, Sieleznieff I, Bertrand M, Marchal F, Dubois A, Pocard M, Rullier A, Smith D, Frulio N, Frison E, Denost Q. Organ preservation with chemoradiotherapy plus local excision for rectal cancer: 5-year results of the GRECCAR 2 randomised trial. Lancet Gastroenterol Hepatol. 2020 May;5(5):465-474. doi: 10.1016/S2468-1253(19)30410-8. Epub 2020 Feb 7. PMID 32043980
- [Background] Bach SP, Gilbert A, Brock K, Korsgen S, Geh I, Hill J, Gill T, Hainsworth P, Tutton MG, Khan J, Robinson J, Steward M, Cunningham C, Levy B, Beveridge A, Handley K, Kaur M, Marchevsky N, Magill L, Russell A, Quirke P, West NP, Sebag-Montefiore D; TREC collaborators. Radical surgery versus organ preservation via short-course radiotherapy followed by transanal endoscopic microsurgery for early-stage rectal cancer (TREC): a randomised, open-label feasibility study. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):92-105. doi: 10.1016/S2468-1253(20)30333-2. Epub 2020 Dec 11. PMID 33308452
- [Background] Brachet S, Meillat H, Chanez B, Ratone JP, Brunelle S, Tyran M, Poizat F, de Chaisemartin C, Lelong B. Case-Matched Comparison of Functional and Quality of Life Outcomes of Local Excision and Total Mesorectal Excision Following Chemoradiotherapy for Rectal Cancer. Dis Colon Rectum. 2022 Dec 1;65(12):1464-1474. doi: 10.1097/DCR.0000000000002384. Epub 2022 Jul 27. PMID 35913830
- [Background] Buess G, Theiss R, Hutterer F, Pichlmaier H, Pelz C, Holfeld T, Said S, Isselhard W. [Transanal endoscopic surgery of the rectum - testing a new method in animal experiments]. Leber Magen Darm. 1983 Mar;13(2):73-7. German. PMID 6621245
- [Background] Rutter MD, Brookes M, Lee TJ, Rogers P, Sharp L. Impact of the COVID-19 pandemic on UK endoscopic activity and cancer detection: a National Endoscopy Database Analysis. Gut. 2021 Mar;70(3):537-543. doi: 10.1136/gutjnl-2020-322179. Epub 2020 Jul 20. PMID 32690602
- [Result] Lewis J, Askari A, Mehta A, Razak Y, Patel P, Misra R, Tilney H, Ahmed T, Ahmed M, Syeed A, Camilleri-Brennan J, Nicholls RJ, Kinross JM. A novel digital rectoscope for the triage of lower gastrointestinal symptoms in primary care: a prospective multicentre feasibility study. BJGP Open. 2022 Sep 28;6(3):BJGPO.2022.0036. doi: 10.3399/BJGPO.2022.0036. Print 2022 Sep. PMID 35728817